CLINICAL TRIAL: NCT02255734
Title: Bioequivalence of Two Formulations of Acyclovir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YSP-REH3002-01
Record Dates: First submitted 2014-05-14; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zovirax (Active Comparator)
  Interventions: Drug: Acyclovir
- Virless (Experimental)
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
Bioequivalence of two formulations of Acyclovir (Acyclovir Lyophilized I.V. infusion 250mg) after Intravenous Infusion in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects between 20 to 45 years of age
* Body weight within 80 to 120 percentages of ideal body weight and higher than or equal to 50 kg for male subjects and 45 kg for female subjects
* Acceptable medical history and physical examination including no particular clinically significant abnormality in x-ray and ECG results within six months prior to period I dosing.no particular clinical significance in general disease history within two months prior to period I dosing
* Acceptable vital signs within normal limits or considered by the investigator or physician to be of no clinical significance at screening, which includes pulse rate, blood pressure and body temperature
* Acceptable clinical chemistry determinations within normal limits or considered by the investigator or physician to be of no clinical significance within two months prior to Period I dosing, which includes AST , ALT ,GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol and triglyceride
* Acceptable hematology within normal range or considered by the investigator or physician to be of no clinical significance within two months prior to Period I dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets
* Acceptable urinalysis within normal limits or considered by the investigator or physician to be of no clinical significance within two months prior to Period I dosing, which includes pH, blood, glucose, ketones, bilirubin and protein
* Female subjects of childbearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigators or surgically sterile bilateral tubal ligation, bilateral oophorectomy or hysterectomy performed on the subject
* Have signed the written informed consent to participate in the study

Exclusion Criteria:

* A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic systems or psychiatric disease as determined by the clinical investigator
* A clinically significant illness or surgery within four weeks prior to Period I dosing as determined by the investigator
* History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years
* History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant
* Known or suspected history of drug abuse within lifetime as judged by the investigator
* History of alcohol addiction or abuse within last five years as judged by the investigator
* History of allergic responses to acyclovir, valacyclovir or any other related drugs
* Evidence of chronic or acute infectious diseases
* Female subjects demonstrating a positive urine pregnancy screen prior to the study
* Female subjects who are currently breastfeeding
* Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to Period I dosing. Examples of inducers include. piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine
* Taking any prescription medications within four weeks or any nonprescription medications excluding flu vaccination within two weeks prior to Period I dosing

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentration | Day 1, Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yen Chen, M.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan